CLINICAL TRIAL: NCT05813730
Title: Definition of Urinary Creatinine Excretion Time in the Neonatal Period, in Full Term Newborns : a Prospective Monocentric Study
Brief Title: Urinary Creatinine Excretion Time in the Neonatal Period
Acronym: C-Rex
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jean-Michel HASCOET, Professor, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RIPH 3 / 2022-A02613-40
Record Dates: First submitted 2023-03-20; First posted 2023-04-14 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Renal Function
Keywords: Newborn; Renal Function; Physiology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy neonates (Other): A single arm evaluating creatinine renal excretion in healthy neonates' urine
  Interventions: Other: urinary creatinine excretion measurement

INTERVENTIONS:
Other: urinary creatinine excretion measurement — Urine samples will be collected up to 6 times a day from birth until discharge from the maternity hospital, to analyze the kinetics of creatinuria.

SUMMARY:
Newborn's renal function is difficult to assess and its physiology during the first days of life is still incompletely known. Studies suggest that the newborn almost completely reabsorbs creatinine during the first 48 to 72 hours of life, while at the same time it continues to produce its own creatinine. Therefore, the initial stock of creatinine at birth still increases through this production and the non or weak clearance. A better knowledge of renal physiopathology in newborns would allow to improve the therapeutic management of the infants, particularly in case of potential nephrotoxicity. No study has attempted to assess the increase in urinary creatinine excretion in neonates from a given time.

Objectives: To show when urinary creatinine excretion in newborns is efficient. Results: this study mightr show an inflection point in urinary creatinine excretion illustrating the postnatal age when renal function becomes efficient.

ELIGIBILITY:
Inclusion Criteria:

* All full-term newborns (37WA or more)
* From a physiological and spontaneous pregnancy
* Good neonatal adaptation (Apgar 7 at 5 minutes of life)
* Eutrophic (weight > 10th percentile and < 90th percentile)

Exclusion Criteria:

* Newborns for whom no urine sample is interpretable
* Those with a significant clinical-biological anomaly
* Neonates with hemodynamic disorders such as low blood pressure (median < gestational age) or hypovolemia (shock, signs of dehydration, need for volume expansion) during the first 3 days of life

Max Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Longitudinal changes in urinary creatinine excretion in newborns | Longitudinal changes of collected samples from birth until discharge from the maternity hospital (i.e. from birth up to 72 hours postnatal age)
  Urine samples will be collected at each diaper change from birth until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie LAMIREAU, Principal Investigator — CHRU Nancy
Locations (1):
- Maternite Regionale Universitaire CHRU NANCY, Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: Undecided